CLINICAL TRIAL: NCT07243457
Title: Incidence Of Urethrocutaneous Fistula Formation In Patients Undergoing Urethroplasty With And Without Stent For Hypospadias
Brief Title: Randomized Trial Of Urethroplasty With Stent Versus Without Stent For Hypospadias
Acronym: UCFStentRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital and Institute of Child Health, Multan (Other Government)
Responsible Party: Principal Investigator, Saira Shafee, Principal Investigator, Children's Hospital and Institute of Child Health, Multan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHM-UCF-Stent-RCT-2025-01; Punjab Health Commission (Other: CHMultan)
Record Dates: First submitted 2025-09-30; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Hypospadias
Keywords: urethroplasty; stent
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Intervention Model Description: Two parallel groups randomized to urethroplasty with stent (Group A) or without stent (Group B); single-center RCT at Children's Hospital Multan.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stented Urethroplasty (Experimental): Standardized urethroplasty performed under general anesthesia with a urethral stent (6-8 Fr nasogastric tube, size by age). Repairs in 3 layers (PDS 6/0 for first/second layers; Polyglactin 5/0 for skin). Stent removed on postoperative day 7; discharge thereafter.
  Interventions: Procedure: Stent urethroplasty
- Stentless Urethroplasty (Active Comparator): Same standardized urethroplasty without a stent; discharge on postoperative day 2.
  Interventions: Procedure: Stentless urethroplasty

INTERVENTIONS:
Procedure: Stent urethroplasty — Urethroplasty with temporary urethral stent (6-8 Fr nasogastric tube) placed intraoperatively and removed on postoperative day 7. Standardized technique: incision after infiltration with 0.5% lignocaine + adrenaline (1:200,000; 5-7 mg/kg), 3-layer repair (PDS 6/0 for first and second layers-interrupted then continuous; Polyglactin 5/0 interrupted for skin). Routine postoperative antibiotics and analgesia. Applies to Arm(s): Stent Urethroplasty (Group A).
  Arms: Stented Urethroplasty
Procedure: Stentless urethroplasty — Urethroplasty without urethral stent using the same standardized operative technique and peri-operative care; planned discharge on postoperative day 2. Applies to Arm(s): Stentless Urethroplasty (Group B).
  Arms: Stentless Urethroplasty

SUMMARY:
Hypospadias is a birth condition in which the urine opening is on the underside of the penis. Surgery (urethroplasty) is the standard treatment. Surgeons sometimes leave a small tube ("stent") inside the new urine passage after surgery, but it is unclear whether using a stent affects the risk of a common complication called a urethrocutaneous fistula (a small leak from the new urethra to the skin).

This study will compare two routine surgical approaches for boys 1-12 years old with distal or mid-penile hypospadias who need urethroplasty: (1) surgery with a temporary stent and (2) surgery without a stent. Children will be randomly assigned to one of the two groups. All surgeries will be performed by a consultant pediatric surgeon using a standardized technique, and all children will receive usual postoperative care.

Families will return for follow-up at 2, 6, and 12 weeks after surgery. At these visits, the team will check for fistula using a simple saline test and record any other concerns. We aim to learn which approach leads to fewer complications, less discomfort, and fewer additional procedures for children undergoing hypospadias repair.

DETAILED DESCRIPTION:
Objective. To compare the incidence of urethrocutaneous fistula (UCF) after hypospadias urethroplasty performed with versus without a postoperative urethral stent. Primary endpoint: UCF at 12 weeks post-operation, defined by saline injection into the neourethra with proximal compression; visible saline spillage between two points is counted as positive.

Design and Setting. Single-center, randomized controlled trial at the Department of Pediatric Surgery, Children's Hospital Multan. Duration: 6 months from synopsis approval. Target sample size: 110 (power 80%, two-proportion test; expected UCF 13.3% with stent vs 33.3% without stent; α=0.05). Allocation by sealed opaque-envelope lottery to two parallel groups.

Participants. Inclusion: boys aged 1-12 years with distal or mid-penile hypospadias scheduled for urethroplasty. Exclusion: prior failed urethroplasty or planned staged repair. Written informed consent from parents/guardians.

Interventions.

Group A (Stent urethroplasty): Standardized urethroplasty with a 6-8 Fr nasogastric tube as temporary stent (size by age). Stent removed on postoperative day 7; discharge thereafter.

Group B (Stentless urethroplasty): Standardized urethroplasty without stent; discharge on postoperative day 2.

All operations under general anesthesia by a consultant pediatric surgeon. Hemostasis with lignocaine 0.5% + adrenaline 1:200,000 (5-7 mg/kg). Repairs in 3 layers (PDS 6/0 first & second layers-interrupted then continuous; skin closure with Polyglactin 5/0 interrupted). Standard postoperative antibiotics and analgesia for both groups.

Follow-up and Assessments. Clinic visits at 2, 6, and 12 weeks. Primary outcome (UCF) assessed with the protocolized saline test; secondary observations include general recovery and any additional interventions. Data captured on a predefined proforma.

Statistical Analysis. Data analyzed in SPSS v23. Normality of numeric variables (e.g., age) by Shapiro-Wilk; age summarized as mean±SD. Categorical variables (site of hypospadias; UCF yes/no) as frequencies/percentages. Primary comparison between groups by chi-square (p<0.05 significant). Stratified analyses by age and hypospadias location with post-stratification chi-square (p<0.05).

Rationale and Significance. Prior comparative studies report differing UCF rates with versus without stents; this trial is designed to provide clearer evidence to guide routine practice, potentially reducing complications, discomfort, and healthcare costs for children undergoing hypospadias repair.

ELIGIBILITY:
Inclusion Criteria: Boys aged 1-12 years

1. Distal or mid-penile hypospadias planned for urethroplasty
2. Parent/guardian provides written informed consent

Exclusion Criteria: Previous failed urethroplasty

1. Planned staged repair

Ages: 1 Year to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2025-05-25 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Urethrocutaneous Fistula at 12 Weeks After Urethroplasty | twelve weeks post operation
  Urethrocutaneous fistula (UCF) will be determined by injecting normal saline under pressure into the terminal neourethra while compressing the penile base; visible saline spillage between two points is counted as positive. Outcome is the proportion of participants with UCF in each arm (stent vs stentless). Assessments occur at routine follow-ups (2, 6, and 12 weeks), with the primary analysis at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Saira Shafee, MBBS, Principal Investigator — Children's Hospital and Institute of Child Health, Multan
Locations (1):
- children Hospital Multan, Multan Khurd, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Demirbilek S, Atayurt HF. One-stage hypospadias repair with stent or suprapubic diversion: which is better? J Pediatr Surg. 1997 Dec;32(12):1711-2. doi: 10.1016/s0022-3468(97)90511-x. PMID 9434004
- [Result] Buson H, Smiley D, Reinberg Y, Gonzalez R. Distal hypospadias repair without stents: is it better? J Urol. 1994 Apr;151(4):1059-60. doi: 10.1016/s0022-5347(17)35180-7. PMID 8126792